CLINICAL TRIAL: NCT06121167
Title: To Examine Whether Urinary Partial Oxygen Pressure Measurements Are Indicative of the Postoperative Occurrence of Acute Kidney Injury (AKI) in Individuals Who Have Undergone Liver Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Murat Bıçakcıoğlu, Asistant prof, Inonu University
Other Study IDs: MB1
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injrury; liver transplantation; urine partial oxygen pressure
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: patients with acute kidney injury
  Interventions: Diagnostic Test: urinary partial oxygen pressure
- control group: patients who do not develop acute kidney injury
  Interventions: Diagnostic Test: urinary partial oxygen pressure

INTERVENTIONS:
Diagnostic Test: urinary partial oxygen pressure — arterial blood gas

SUMMARY:
Postoperative acute kidney injury (AKI) is a frequent occurrence among liver transplant recipients and results in considerable mortality and morbidity. The delayed increase in plasma creatinine levels and its susceptibility to external influences, which are utilized in the current diagnostic criteria for AKI, contribute to diagnostic delays. Therefore, numerous biomarkers, including KIM-1, NGAL, TIMP-2, and CYSTATIN C in plasma, along with urine partial oxygen pressure levels and NGAL, are currently under examination to identify acute kidney injury at its early stage. It is well-established that the renal medulla is highly susceptible to hypoxia, which may consequently lead to acute kidney injury. A range of studies have also demonstrated that urine partial oxygen pressure is capable of providing valuable insights into the oxygenation state of the renal medulla. Although urine oxygen pressure measurement is not commonly used, unlike blood gas analysis, urine partial oxygen pressure measurement dates back to 1964. Research among cardiopulmonary bypass patients suggests a correlation between urine partial oxygen pressure data and acute kidney injury. Therefore, we hypothesize that monitoring urine partial oxygen pressure levels may offer insight into the development of acute kidney injury in liver transplant recipients.

DETAILED DESCRIPTION:
Ninety-eight participants, aged between 18 and 65 and scheduled for elective liver transplantation, will participate in this study. Participants under the age of 18, those who decline participation, those undergoing transplantation due to fulminant hepatic failure, those who develop hepatic encephalopathy, and patients with hepatorenal or hepatopulmonary syndrome or previous lung and heart disease will not be considered for inclusion. After obtaining ethical approval, the patients will undergo a preanaesthetic examination. Upon admission to the procedure room, standard monitoring for liver transplant recipients will be conducted. Thiopental at a dose of 5-8 mg/kg, fentanyl at 1-2 mcg/kg, lidocaine at 1 mg/kg, and vecuronium at 0 will be administered. Technical term abbreviations will be explained upon first use. The structure and language used in the text adhere to the principles of academic writing. Consistent citation and formatting features will be followed. Grammatical correctness, clear language, and logical progression of information will be prioritised. Biased language and ornamental language will be avoided. Anaesthesia will be administered at a dosage of 1 mg/kg. Following proper anaesthetic depth, intubation will take place. A urine sample (T0) and arterial blood gas will be obtained from the urinary catheter via syringe, with the aid of a blood gas analyser device before the surgical procedure. Partial pressure of oxygen will also be recorded. Before the patient departs the operating theatre, a urine sample and arterial blood gas (T1) will be retaken with a syringe and the partial oxygen level measured. Throughout the operation, data on haemodynamics, respiration, routine lab results, hourly urine output, as well as diuretic and vasopressor requirements (if applicable), will be captured. The total duration of the operation will be recorded at its conclusion. At the 18th hour post-op, a urine and arterial blood sample (T2) will be taken to measure partial oxygen pressure levels. Additionally, the NGAL level in plasma will be studied. At the 48th hour postoperative, partial oxygen pressure levels in urine and arterial blood (T3) will be measured, and the obtained data will be recorded. Please adhere to the standardised technical terminology when referencing these measurements. The quantity of urine output per hour, CSDGO score, requirement for vasopressors, diuretics, RRT, mechanical ventilation, and any subsequent complications will be documented in the intensive care unit postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18 and 65 years
* elective liver transplantation

Exclusion Criteria:

* Patients who do not want to participate in the study,
* patients who will be transplanted due to fulminant hepatic failure,
* patients with hepatic encephalopathy,
* patients with hepatorenal or hepatopulmonary syndrome,
* patients with previous lung
* heart disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: liver transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2024-03-06 (Estimated); Primary Completion 2024-05-10 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
acute kidney injury | first 7 days
  whether urinary oxygen partial pressure can predict acute kidney injury

SECONDARY OUTCOMES:
mortality | 28. days
  death rate

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tosun M, Ulugol H, Aksu U, Toraman F. Can Partial Oxygen Pressure of Urine be an Indicator for Tissue Perfusion? Turk J Anaesthesiol Reanim. 2019 Jun;47(3):187-191. doi: 10.5152/TJAR.2019.89083. Epub 2019 Jan 29. PMID 31183464
- [Background] Silverton NA, Lofgren LR, Hall IE, Stoddard GJ, Melendez NP, Van Tienderen M, Shumway S, Stringer BJ, Kang WS, Lybbert C, Kuck K. Noninvasive Urine Oxygen Monitoring and the Risk of Acute Kidney Injury in Cardiac Surgery. Anesthesiology. 2021 Sep 1;135(3):406-418. doi: 10.1097/ALN.0000000000003663. PMID 34329393
- [Result] Stafford-Smith M. Could Trended Oxygen Partial Pressure in the Urine Be the "ST Segment" Kidney Monitor We've Been Looking For? Anesthesiology. 2021 Sep 1;135(3):380-381. doi: 10.1097/ALN.0000000000003869. No abstract available. PMID 34329391